CLINICAL TRIAL: NCT04334668
Title: Oral Sodium to Preserve Renal EfficiencY in Acute Heart Failure (OSPREY-AHF)
Brief Title: Oral Sodium to Preserve Renal EfficiencY in Acute Heart Failure
Acronym: OSPREY-AHF
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The Cleveland Clinic (Other)
Responsible Party: Principal Investigator, Wilson Tang, Principal Investigator, Staff Cardovascular & Metabolic Sciences and Cardiovascular Medicine, The Cleveland Clinic, The Cleveland Clinic
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: 20-183
Record Dates: First submitted 2020-04-01; First posted 2020-04-06 (Actual); Results first posted 2024-03-12 (Actual); Last update posted 2025-05-04 (Actual); Status verified 2025-04

CONDITIONS: Volume Overload
MeSH Terms: conditions — Edema | interventions — Sodium Chloride

STUDY DESIGN:
Intervention Model Description: Heart Failure patients hospitalized for diuresis
Who Masked: Participant, Care Provider
Masking Description: This is a double blind study. Subjects will be randomized to Sodium Chloride tablets and Placebos and picked up from pharmacy.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Oral Sodium Chloride (Active Comparator): Subject will be given 2 grams of oral sodium chloride three times daily with meals for approximately 4 days
  Interventions: Dietary Supplement: Oral Sodium Chloride
- Placebo (Placebo Comparator): Subject will be given a placebo orally three times daily with meals for approximately 4 days
  Interventions: Other: Placebo

INTERVENTIONS:
Dietary Supplement: Oral Sodium Chloride — Subjects will be randomized to receive 2 grams oral Sodium Chloride three times daily with meals for approximately 4 days
  Arms: Oral Sodium Chloride
Other: Placebo — Subjects will be randomized to receive a placebo three times daily with meals for approximately 4 days.
  Arms: Placebo

SUMMARY:
The investigators are proposing a prospective, randomized, double blinded, placebo-controlled single center study evaluating the role of co-administration of oral sodium chloride (NaCl) with intravenous diuretics in patients hospitalized with acute decompensated heart failure. The investigators are approaching this study with the hypothesis that the use of oral sodium chloride leads to improved effective diuresis (as measured by weight loss) and renal function as compared to placebo in patients hospitalized with acute decompensated heart failure undergoing aggressive intravenous diuretic therapy.

DETAILED DESCRIPTION:
Dietary sodium restriction is a common therapeutic intervention in the management of patients hospitalized with decompensated heart failure. This is despite limited supportive data and inconsistent society guidelines.1-3 Randomized clinical trial data has shown that dietary sodium restriction in patients hospitalized with heart failure was not associated with differences in weight, clinical congestion, time to clinical stability but was associated with increased thirst.4 Numerous studies demonstrate that sodium restriction is associated with increased Renin-Angiotensin-Aldosterone System (RAAS) activation as well as increases in inflammatory markers.5,6 These findings challenge of the role of sodium restriction in hospital management of heart failure and have lead to trials that consider a therapeutic role of providing sodium to patients with acute heart failure for its effect in attenuating neurohormonal activation during aggressive diuresis. A central example is the SMAC-HF study from Italy, which showed that in 1771 patients with acute New York Heart Association (NYHA) class IV heart failure, the addition of hypertonic saline (150ml of 1.4%-4.6% NaCl twice a day in addition to diet liberalization led to statistically significant increased urine output and weight loss in addition to reductions in creatinine, length of stay, mortality and readmissions.7 These findings are controversial but similarly favorable results with the use of hypertonic saline in aiding diuresis have been seen in Japan with improved diuresis with continuous hypertonic saline infusions.8 Despite these results, use of sodium chloride supplementation in acute heart failure remains limited. This may be because the practice challenges ingrained clinical practice, but a more likely reason is that the manner of sodium chloride delivery in these trials (hypertonic saline) is often reserved for the Intensive Care Unit (ICU) setting and central venous access for delivery. While small volumes of hypertonic saline are likely safe to be administered in a non-ICU setting, the results would be more broadly applicable and utilized if the manner of sodium supplementation did not require intensive monitoring or central venous access, ie oral supplementation. Therefore, the purpose of the "Oral Sodium to Preserve Renal EfficiencY in Acute Heart Failure" (OSPREY-AHF) is to evaluate the efficacy and safety of oral sodium chloride supplementation compared to placebo in patients with acute decompensated heart failure. While the investigators are specifically interested in sodium chloride and its hypothesized role in attenuating a neurohormonally mediated diuretic resistance commonly seen in patients requiring high dose diuretic therapy, the investigators also intend that by focusing on oral sodium chloride supplementation the investigators may clarify the role of dietary sodium restriction in hospitalized patients with acute heart failure.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years old AND
* Admitted to cardiology floor (non-ICU) with primary diagnosis of decompensated heart failure AND
* NT-proBNP >1000 ng/L AND
* Initiation of continuous furosemide infusion at a rate of 10 mg/hr or higher

Exclusion Criteria:

* Serum sodium (Na+) level less than 120 or greater than 145.
* Average Systolic Blood Pressure >180 mmHg or Diastolic Blood Pressure >100 mmHg over past 24 hours.
* Anticipated length of stay less than 72 hours.
* Use of vasopressin antagonist
* Current use of sodium chloride tablets
* Active diagnosis of diabetes insipidus
* Inability to tolerate oral diet or swallow pills
* Presence of malabsorptive gastrointestinal disorder (Crohn's disease, short gut syndrome)
* The use of iodinated radiocontrast material in the past 72 hours or anticipated use of intravenous contrast during the current hospitalization
* Admission with intention to transplant or implant permanent Ventricular Assistive Device
* Use of intravenous inotropes, vasopressors or vasodilators at enrollment
* A baseline estimated glomerular filtration rate <15 mL/min/1.73m² according to the Chronic Kidney Disease Epidemiology Collaboration (CKD-EPI) formula at the moment of inclusion
* Use of renal replacement therapy at time of enrollment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 67 (Actual)
Dates: Start 2020-05-20 (Actual); Primary Completion 2022-06-01 (Actual); Study Completion 2026-06-01 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: W. H. Wilson Tang, MD, Principal Investigator — The Cleveland Clinic; Robert A Montgomery, MD, Principal Investigator — The Cleveland Clinic
Locations (1):
- Cleveland Clinic, Cleveland, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Yancy CW, Jessup M, Bozkurt B, Butler J, Casey DE Jr, Drazner MH, Fonarow GC, Geraci SA, Horwich T, Januzzi JL, Johnson MR, Kasper EK, Levy WC, Masoudi FA, McBride PE, McMurray JJ, Mitchell JE, Peterson PN, Riegel B, Sam F, Stevenson LW, Tang WH, Tsai EJ, Wilkoff BL; American College of Cardiology Foundation; American Heart Association Task Force on Practice Guidelines. 2013 ACCF/AHA guideline for the management of heart failure: a report of the American College of Cardiology Foundation/American Heart Association Task Force on Practice Guidelines. J Am Coll Cardiol. 2013 Oct 15;62(16):e147-239. doi: 10.1016/j.jacc.2013.05.019. Epub 2013 Jun 5. No abstract available. PMID 23747642
- [Background] Heart Failure Society of America; Lindenfeld J, Albert NM, Boehmer JP, Collins SP, Ezekowitz JA, Givertz MM, Katz SD, Klapholz M, Moser DK, Rogers JG, Starling RC, Stevenson WG, Tang WH, Teerlink JR, Walsh MN. HFSA 2010 Comprehensive Heart Failure Practice Guideline. J Card Fail. 2010 Jun;16(6):e1-194. doi: 10.1016/j.cardfail.2010.04.004. PMID 20610207
- [Background] McMurray JJ, Adamopoulos S, Anker SD, Auricchio A, Bohm M, Dickstein K, Falk V, Filippatos G, Fonseca C, Gomez-Sanchez MA, Jaarsma T, Kober L, Lip GY, Maggioni AP, Parkhomenko A, Pieske BM, Popescu BA, Ronnevik PK, Rutten FH, Schwitter J, Seferovic P, Stepinska J, Trindade PT, Voors AA, Zannad F, Zeiher A; ESC Committee for Practice Guidelines. ESC Guidelines for the diagnosis and treatment of acute and chronic heart failure 2012: The Task Force for the Diagnosis and Treatment of Acute and Chronic Heart Failure 2012 of the European Society of Cardiology. Developed in collaboration with the Heart Failure Association (HFA) of the ESC. Eur Heart J. 2012 Jul;33(14):1787-847. doi: 10.1093/eurheartj/ehs104. Epub 2012 May 19. No abstract available. PMID 22611136
- [Background] Aliti GB, Rabelo ER, Clausell N, Rohde LE, Biolo A, Beck-da-Silva L. Aggressive fluid and sodium restriction in acute decompensated heart failure: a randomized clinical trial. JAMA Intern Med. 2013 Jun 24;173(12):1058-64. doi: 10.1001/jamainternmed.2013.552. PMID 23689381
- [Background] Graudal NA, Hubeck-Graudal T, Jurgens G. Effects of low-sodium diet vs. high-sodium diet on blood pressure, renin, aldosterone, catecholamines, cholesterol, and triglyceride (Cochrane Review). Am J Hypertens. 2012 Jan;25(1):1-15. doi: 10.1038/ajh.2011.210. Epub 2011 Nov 9. PMID 22068710
- [Background] Parrinello G, Di Pasquale P, Licata G, Torres D, Giammanco M, Fasullo S, Mezzero M, Paterna S. Long-term effects of dietary sodium intake on cytokines and neurohormonal activation in patients with recently compensated congestive heart failure. J Card Fail. 2009 Dec;15(10):864-73. doi: 10.1016/j.cardfail.2009.06.002. PMID 19944363
- [Background] Paterna S, Fasullo S, Parrinello G, Cannizzaro S, Basile I, Vitrano G, Terrazzino G, Maringhini G, Ganci F, Scalzo S, Sarullo FM, Cice G, Di Pasquale P. Short-term effects of hypertonic saline solution in acute heart failure and long-term effects of a moderate sodium restriction in patients with compensated heart failure with New York Heart Association class III (Class C) (SMAC-HF Study). Am J Med Sci. 2011 Jul;342(1):27-37. doi: 10.1097/MAJ.0b013e31820f10ad. PMID 21701268
- [Background] Okuhara Y, Hirotani S, Naito Y, Nakabo A, Iwasaku T, Eguchi A, Morisawa D, Ando T, Sawada H, Manabe E, Masuyama T. Intravenous salt supplementation with low-dose furosemide for treatment of acute decompensated heart failure. J Card Fail. 2014 May;20(5):295-301. doi: 10.1016/j.cardfail.2014.01.012. Epub 2014 Jan 22. PMID 24462960
- [Derived] Montgomery RA, Mauch J, Sankar P, Martyn T, Engelman T, Martens P, Faulkenberg K, Menon V, Estep JD, Tang WHW. Oral Sodium to Preserve Renal Efficiency in Acute Heart Failure: A Randomized, Placebo-Controlled, Double-Blind Study. J Card Fail. 2023 Jul;29(7):986-996. doi: 10.1016/j.cardfail.2023.03.018. Epub 2023 Apr 11. PMID 37044281

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Oral Sodium Chloride | Placebo
Started | 34 | 33
Completed | 34 | 31
Not Completed | 0 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Oral Sodium Chloride | Placebo | Total
Number analyzed (Participants) | 34 | 31 | 65
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 10 | 10 | 20
  >=65 years | 24 | 21 | 45
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14 | 11 | 25
  Male | 20 | 20 | 40
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 34 | 31 | 65
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 7 | 2 | 9
  White | 27 | 29 | 56
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 34 | 31 | 65

OUTCOME MEASURES:

1. Primary Outcome: Change in Weight
Description: Measured in kilograms
Time Frame: Baseline to 96 hours
Measure: Mean (Standard Deviation); unit: Kilograms
Arm/Group | Oral Sodium Chloride | Placebo
Number analyzed (Participants) | 34 | 31
Kilograms | -3.9 (4.3) | -4.6 (4.2)

2. Primary Outcome: Change in Creatinine
Description: Measured in milliequivalents per Liter
Time Frame: Baseline to 96 hours
Measure: Mean (Standard Deviation); unit: mEq/L
Arm/Group | Oral Sodium Chloride | Placebo
Number analyzed (Participants) | 34 | 31
mEq/L | 0.038 (0.39) | 0.15 (0.44)

ADVERSE EVENTS:
Time Frame: Enrollment to 90 days post enrollment
Arm/Group | Oral Sodium Chloride | Placebo
All-Cause Mortality (participants affected / at risk) | 3/34 | 3/31
Serious Adverse Events (participants affected / at risk) | 7/34 | 7/31
Other Adverse Events (participants affected / at risk) | 4/34 | 4/31
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Oral Sodium Chloride (N=34) | Placebo (N=31)
Worsening Renal Function (Renal and urinary disorders) | 0 (0) | 1 (1) — >48 hours after study medication completion subject had worsening Renal Function, Right Heart Catheterization showed low output. Transferred to ICU for vasodilation.
Low output and elevated filling pressure (Cardiac disorders) | 1 (1) | 0 (0) — Low cardiac output & elevated filling pressures found during right heart catherization. Transferred to ICU for swan guided afterload optimization. Study drug discontinued 24 hours prior to discontinuation of IV diuretic.
Hypokalemia (General disorders) | 0 (0) | 1 (1) — 35 days after receiving final study medication patient readmitted with hypokalemia & ICD shock aborted cardiac arrest from VF. Patient had a history of ICD shocks. Incident & hypokalemia occurred after receiving metolazone (unrelated to the study).
Readmission for weight gain (General disorders) | 1 (1) | 0 (0) — Readmission with weight gain and lower extremity swelling secondary to recurrent heart failure. Diuresed with lasix and discharged 4 days later.
ICU transfer (Cardiac disorders) | 0 (0) | 1 (1) — Underwent Right Heart Catheterization which revealed markedly elevated filling pressures and low cardiac index. Transferred to CICU. Hemodynamics improved with sodium nitroprusside.
Readmitted (General disorders) | 0 (0) | 1 (1) — Hemoglobin dropped to 5.6, down from 8. Received 2 units of blood with appropriate subsequent rise in hemoglobin.
VF arrest (Cardiac disorders) | 0 (0) | 1 (1) — Passed away after a VF arrest. Developed pulseless VT in the setting of un-revascularized coronary disease and severe biventricular cardiomyopathy.
Readmission (General disorders) | 1 (1) | 0 (0) — Patient readmitted with high blood pressure, diffuse joint pain, and compensated heart failure. Rheumatology felt presentation was consistent with either reactive arthritis or hydralazine induced arthralgias, unrelated to the study.
COVID 19 infection (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) — Readmission for shortness of breath. Died during admission from COVID-19 infection. Death and readmission not related to study drug.
ICU transfer (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) — Patient transferred to ICU for hematemesis and underwent squamous carcinoma resection. Patient transitioned to DNRCC and died of respiratory failure in the setting of post-operative complications from bladder malignancy surgery.
Leukocytosis and worsening renal function (General disorders) | 1 (1) | 0 (0) — Readmitted for fluid overload. Developed altered mental status related to leukocytosis & worsening renal function. Dialysis didn't improve mental status. Made DNR/DNI & died on day of transfer to hospice. Only 1 dose of study medication taken.
Respiratory decompensation (General disorders) | 0 (0) | 1 (1) — ICU transfer and subsequent death related to respiratory decompensation from aspiration & pulmonary infection. Acute Kidney Injury and worsening respiratory function followed. Unrelated to study.
Readmission (General disorders) | 0 (0) | 1 (1) — Readmission with worsening renal function and heart failure. Occurrence >3weeks after study medication, unrelated to study.
Uncontrolled dyspnea (General disorders) | 1 (1) | 0 (0) — Readmitted with neutropenic fever related to leukemia. Admitted to hospice for uncontrolled dyspnea and died. Unrelated to study medication
ICU transfer (General disorders) | 0 (0) | 1 (1) — Creatinine increased from 1.01 on admission to 1.98 on study day one. Transferred to ICU. Subsequent Right Heart Catheterization showed elevated biventricular filling pressures & normal cardiac index. Unlikely to be related to study.
ICU (General disorders) | 1 (1) | 0 (0) — During the study a routine clinical Right Heart Catheterization was performed to assess volume status. Patient transferred to CICU due to elevated filling pressures and low output therapy. Cardiac index normalized with nitroprusside therapy.
Increase in creatinine (Renal and urinary disorders) | 1 (1) | 0 (0) — Creatinine increased from 2.6 at End of Study visit to 3.19 eight days post study. Dialysis started and renal function improved. Unlikely to be study related
ICU (Cardiac disorders) | 0 (0) | 1 (1) — Transferred to ICU 5 days post study. Pulmonary Artery catheter numbers showed Pulmonary Capillary Wedge Pressure 34 and Cardiac Index 1.96. Accepted for LVAD at a later date.
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Oral Sodium Chloride (N=34) | Placebo (N=31)
Gout Flare up (General disorders) | 0 (0) | 1 (1) — Gout flare up, likely due to diuretic use and unlikely related to study medication.
hypokalemia (General disorders) | 0 (0) | 1 (1) — Hypokalemia (K3.1), required holding of lasix. Hypokalemia is a common side effect of metolazone. Unable to rule out study medication as cause.
Hypokalemia, VF arrest (General disorders) | 0 (0) | 1 (1) — Hypokalemia, VF arrest, ICD shock aborted cardiac arrest. Patient history of ICD shocks. Incident and hypokalemia occurred after receiving metolazone. Can't rule out study medication as the cause.
Transferred to ICU (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) — Transferred to ICU for lethargy & hypoxia. Treated for aspiration pneumonia/pneumonitis on top of baseline pulmonary congestion. Unlikely to be related to study medication.
Hyponatremia (General disorders) | 1 (1) | 0 (0) — 2 days after study medication finished patient developed hyponatremia. Sodium level decreased from 131 to 125.
Nausea (Gastrointestinal disorders) | 0 (0) | 1 (1) — 1 dose of study medication held due to patient nausea
Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0) — Patient developed nausea after 1st dose of study medication
Nausea/Vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0) — Patient stated they threw up the first dose of study medication and didn't take any more.

LIMITATIONS AND CAVEATS:
Limitations: single center trial, small sample size, heterogeneous baseline characteristics & degree of congestion, only powered for short term effects of NaCl supplementation, not powered for noninferiority analysis for change in weight, extra NaCl not continued after IV diuresis stopped, underpowered to fully assess significance of NaCl on safety, only spot urine collected (no 24-hour urine) & only 48 patients provided samples for serum biomarker analysis.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-03-12): https://cdn.clinicaltrials.gov/large-docs/68/NCT04334668/Prot_SAP_000.pdf